CLINICAL TRIAL: NCT02874573
Title: A Randomized Controlled Trial of Adjunctive Tocilizumab in Schizophrenia
Brief Title: Tocilizumab in Schizophrenia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brian Miller (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Brian Miller, Associate Professor, Augusta University
Organization: Augusta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 944642
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Inflammation; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Inflammation | interventions — tocilizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Active Comparator): Subjects in the tocilizumab group will receive a 4 mg/kg infusion at baseline, and weeks 4 and 8, as per the recommended starting dosing for rheumatoid arthritis
  Interventions: Drug: Tocilizumab
- Control Group (Placebo Comparator): Subjects in the placebo group will receive an infusion of normal saline (with the same packaging and volume as the tocilizumab group) at baseline, and weeks 4 and 8.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tocilizumab — Investigational agent
  Other Names: Actemra
  Arms: Treatment Group
Drug: Normal saline — Placebo
  Other Names: 0.9% NS
  Arms: Control Group

SUMMARY:
This study is a Phase 1 clinical trial to determine the safety, tolerability, and efficacy of Tocilizumab (Actemra) as an adjunct to antipsychotic medications in stable outpatients with schizophrenia. Tocilizumab (structural formula C6428H9976N1720O2018S42) is a recombinant humanized anti-human interleukin-6 (IL-6) receptor monoclonal antibody of the immunoglobulin G1 (IgG1) subclass. Tocilizumab is formulated as a concentrate for solution for infusion, and will be administered by intravenous infusion.

The investigators propose a 12-week randomized controlled trial of tocilizumab, given in adjunct to antipsychotics, in N=20 stable outpatients with schizophrenia or schizoaffective disorder and evidence of increased inflammation in the peripheral blood (high-sensitivity C-reactive protein [hsCRP]>0.5 mg/dL). The investigators hypothesize that adjunctive treatment with tocilizumab will be associated with significant improvement in cognition compared to placebo in patients with schizophrenia, and baseline IL-6 levels are higher in tocilizumab-treated responders versus non-responders, and there will be greater decreases in hsCRP from baseline to week 12 in tocilizumab-versus placebo-treated responders, with response defined as ≥0.5 standard deviation (SD) improvement in cognition. Tocilizumab is administered as an intravenous infusion every 4 weeks. Following a screening evaluation, participants will receive three infusions of siltuximab, one at baseline, another at week 4 of the study, and another at week 8. The investigators will measure changes in cognitive function and symptoms over a 12-week period. Complementing previous positive clinical trials of non-steroidal anti-inflammatory drugs, this would be a "proof-of-concept" study that targeting specific cytokines is a viable treatment for schizophrenia.

Interleukin 6 and its receptor were discovered and cloned at Osaka University, Japan, by Tadamitsu Kishimoto in the 1980s. In 1997, Chugai Pharmaceuticals began the clinical development of tocilizumab for the treatment of rheumatoid arthritis. Clinical studies for Castleman's disease and systemic juvenile idiopathic arthritis started in 2001 and 2002, respectively. Hoffmann-La Roche co-developed the drug due to a license agreement in 2003.

On 11 January 2010, Tocilizumab was approved by the U.S. Food and Drug Administration (US FDA) as Actemra for the treatment of rheumatoid arthritis. The FDA approved tocilizumab for the treatment of systemic juvenile idiopathic arthritis for children from two years of age in April 2011.

DETAILED DESCRIPTION:
A pathophysiological role for inflammation in schizophrenia has been one of the more enduring findings in the field. Recently, increased understanding of complex interactions between inflammation and the brain in other chronic diseases has better informed this relationship in schizophrenia. Several trials have found that treatment with non-steroidal anti-inflammatory drugs (NSAIDs), in adjunct to antipsychotics, was associated with significant improvement in psychopathology in schizophrenia. Cytokines are key regulators of inflammation that exert effects in the periphery and the brain. Serum cytokine levels predicted response in two studies, and another study found a trend for improved cognition with adjunctive NSAID treatment.1 These findings provide important empirical support for a pathophysiological role for inflammation in some patients with schizophrenia. Two important limitations of these trials are that: a) the agents investigated have relevant off-target (i.e., non-immune) effects, and b) evidence of inflammation in the peripheral blood was not an inclusion criterion, which may have decreased the signal-to-noise ratio.

Schizophrenia is associated with impaired cognition, which persists despite current treatments, and is an important determinant of quality of life and overall function. Converging lines of evidence suggest that interleukin-6 (IL-6) is a promising therapeutic target for cognitive impairment in schizophrenia. IL-6 is a cytokine produced by peripheral blood leukocytes, and central nervous system (CNS) microglia and astrocytes. The IL-6 gene is a risk factor for schizophrenia and may impact on serum IL-6 levels. Blood and (cerebrospinal fluid) CSF IL-6 levels are altered in schizophrenia. IL-6 levels are associated with psychopathology3 and cognition in schizophrenia. In populations outside of schizophrenia, higher serum IL-6 levels are associated with poorer cognition. In first-episode and chronic schizophrenia, IL-6 levels are a significant predictor of smaller left hippocampal volume.

Along with our other previous work, our preliminary studies provide strong evidence that IL-6 is a novel therapeutic target for cognitive impairment in schizophrenia, and demonstrate the feasibility of the proposed trial. Briefly, in 64 patients with schizophrenia, we found higher blood IL-6 levels were a significant predictor of greater impairment on the Brief Assessment of Cognition in Schizophrenia (BACS) after controlling for multiple potential confounding factors.5 In an 8-week open-label trial in 6 subjects, tocilizumab (a humanized monoclonal antibody against the IL-6 receptor, approved by the US FDA in 2010 for the treatment of adults with moderately to severely active rheumatoid arthritis (RA) who have had an inadequate response to one or more tumor necrosis factor (TNF)-antagonist therapies, administered as an intravenous infusion every 4 weeks), given in adjunct to antipsychotics, was well tolerated and associated with significant improvement in BACS verbal fluency at 4 weeks, BACS digit symbol coding at 2, 4, and 8 weeks, and BACS composite score at 4 and 8 weeks.10

In the first year following the submission, one clinical trial is planned. The investigators will conduct a 12-week randomized, double-blind, placebo-controlled trial to determine the safety, tolerability, and efficacy of tocilizumab as an adjunct to antipsychotic medications in 20 stable outpatients with schizophrenia.

In our previous trial of Tocilizumab, no clinically significant adverse drug reactions occurred. The risks that have been found in people with rheumatoid arthritis are known, but there may be unknown risks when used in schizophrenia. Clinically significant adverse drug reactions include anaphylaxis (0.4%), infections (0.1-7.8%), intestinal perforation, neutropenia (7.0%), and cardiac failure. Known side effects of tocilizumab that are common include: increase in hepatic enzymes (AST, ALT), hypertension, headache, neutropenia, infusion-related reactions, upper respiratory tract infections, and nasopharyngitis.

Subjects with schizophrenia and schizoaffective disorder will be accessed from outpatient psychiatry clinic at Augusta University or other satellite collaborative sites. The study has 6 visits: screening, baseline, and weeks 2, 4, 8, and 12. Subjects will be randomized equally to either tocilizumab (n=10) or placebo (n=10), in adjunct to their current antipsychotic and other psychotropic medications. Tocilizumab will be obtained from the manufacturer, Genentech, through our hospital pharmacy as per our previous trial. Subjects in the tocilizumab group will receive a 4 mg/kg infusion at baseline, and weeks 4 and 8, as per the recommended starting dosing for rheumatoid arthritis. Subjects in the placebo group will receive an infusion of normal saline (with the same packaging and volume as the tocilizumab group) at baseline, and weeks 4 and 8. We will contact the subjects by phone on days 1 and 7 after each infusion to assess for any infusion-related events. We will assess cognition and psychopathology at baseline, and at weeks 2, 4, 8, and 12. We will also measure a multiplex panel of blood cytokines (including IL-6) at baseline, and at weeks 2m 4, 8, and 12. Patients will be withdrawn if they meet any exclusion criterion at any time point.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* age 18-55
* capable of giving informed consent
* Diagnostic and Statistical Manual of Mental Disorders (DSM)-V diagnosis of schizophrenia or schizoaffective disorder
* stable based on clinical judgment, no psychiatric hospitalizations in past 3 months, and on the same psychotropic medications for >4 weeks
* taking a non-clozapine antipsychotic
* hsCRP >0.3 mg/dL at the screening visit

Exclusion Criteria:

* imminent danger to self/others
* antibiotic use in the past 2 weeks
* current scheduled use of immunomodulatory agents
* history of an immune disorder
* illicit drug use in the past 30 days
* any unstable or untreated medical condition
* history of gastrointestinal ulcers, diverticulitis, malignancy, CNS demyelinating disorder, seizure disorder, or tuberculosis
* low absolute neutrophil (<2000) or platelet (<100,000) count
* abnormal hepatic (AST or ALT >1.5 times the upper limit of normal) or renal (BUN or creatinine>1.5 times the upper limit of normal) function
* any abnormal lab test result judged to be clinically significant
* active, chronic or recurrent infections
* pregnancy
* breast feeding
* female and of child-bearing potential who is not using any contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition | Baseline and 12 weeks
  The Brief Assessment of Cognition in Schizophrenia (BACS) is the metric used to characterize cognition in this study. The BACS consists of 6 subscales: Verbal Memory (range 0-75), Working Memory (range 0-28), Motor Speed (range 0-100), Verbal Fluency (measure is total number of words generated in two 60 second trials), Attention and Processing speed (range 0-110), and Executive Function (range 0-22). For each subscale, higher scores reflect better cognition. For each subscale, a Standard Deviation Score was calculated based on normative data (Keefe et al. Norms and standardization of the Brief Assessment of Cognition in Schizophrenia (BACS). Schizophrenia Research 102 (2008) 108-115). The BACS composite score is calculated as the average Standard Deviation Score of the 6 subscale scores. The change in BACS composite score will be calculated as the BACS composite score at 9 weeks minus the BACS composite score at baseline.

SECONDARY OUTCOMES:
Change in Total Psychotic Symptoms | Baseline and 12 weeks
  The Positive and Negative Symptoms Scale (PANSS) is the metric used to characterize psychotic symptoms in this study. The PANSS consists of 30 items, each scored 1-7. The range for the PANSS total score is 30-210. There are 3 subscales - PANSS positive score (range 7-49), PANSS negative score (range 7-49), and PANSS general score (range 16-112). PANSS total score is the summation of these 3 subscales. Higher values for the total and subscale scores reflect more severe psychopathology. A positive change in PANSS total score reflects an increase in psychopathology. A negative change in PANSS total score reflects a decrease in psychopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Miller, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

REFERENCES:
- [Background] Nitta M, Kishimoto T, Muller N, Weiser M, Davidson M, Kane JM, Correll CU. Adjunctive use of nonsteroidal anti-inflammatory drugs for schizophrenia: a meta-analytic investigation of randomized controlled trials. Schizophr Bull. 2013 Nov;39(6):1230-41. doi: 10.1093/schbul/sbt070. Epub 2013 May 29. PMID 23720576
- [Background] Sasayama D, Wakabayashi C, Hori H, Teraishi T, Hattori K, Ota M, Ishikawa M, Arima K, Higuchi T, Amano N, Kunugi H. Association of plasma IL-6 and soluble IL-6 receptor levels with the Asp358Ala polymorphism of the IL-6 receptor gene in schizophrenic patients. J Psychiatr Res. 2011 Nov;45(11):1439-44. doi: 10.1016/j.jpsychires.2011.06.003. Epub 2011 Jun 22. PMID 21700295
- [Background] Miller BJ, Buckley P, Seabolt W, Mellor A, Kirkpatrick B. Meta-analysis of cytokine alterations in schizophrenia: clinical status and antipsychotic effects. Biol Psychiatry. 2011 Oct 1;70(7):663-71. doi: 10.1016/j.biopsych.2011.04.013. Epub 2011 Jun 8. PMID 21641581
- [Background] Sasayama D, Hattori K, Wakabayashi C, Teraishi T, Hori H, Ota M, Yoshida S, Arima K, Higuchi T, Amano N, Kunugi H. Increased cerebrospinal fluid interleukin-6 levels in patients with schizophrenia and those with major depressive disorder. J Psychiatr Res. 2013 Mar;47(3):401-6. doi: 10.1016/j.jpsychires.2012.12.001. Epub 2013 Jan 3. PMID 23290488
- [Background] Frydecka D, Misiak B, Pawlak-Adamska E, Karabon L, Tomkiewicz A, Sedlaczek P, Kiejna A, Beszlej JA. Interleukin-6: the missing element of the neurocognitive deterioration in schizophrenia? The focus on genetic underpinnings, cognitive impairment and clinical manifestation. Eur Arch Psychiatry Clin Neurosci. 2015 Sep;265(6):449-59. doi: 10.1007/s00406-014-0533-5. Epub 2014 Sep 12. PMID 25214388
- [Background] Miller B, Mellor A, Buckley PF. Interleukin-6 and Cognition in Non-Affective Psychosis. Schizophr Bull 2013; 39: S242-S243.
- [Background] Marsland AL, Petersen KL, Sathanoori R, Muldoon MF, Neumann SA, Ryan C, Flory JD, Manuck SB. Interleukin-6 covaries inversely with cognitive performance among middle-aged community volunteers. Psychosom Med. 2006 Nov-Dec;68(6):895-903. doi: 10.1097/01.psy.0000238451.22174.92. PMID 17132839
- [Background] Kalmady SV, Venkatasubramanian G, Shivakumar V, Gautham S, Subramaniam A, Jose DA, Maitra A, Ravi V, Gangadhar BN. Relationship between Interleukin-6 gene polymorphism and hippocampal volume in antipsychotic-naive schizophrenia: evidence for differential susceptibility? PLoS One. 2014 May 2;9(5):e96021. doi: 10.1371/journal.pone.0096021. eCollection 2014. PMID 24787542
- [Background] Miller BJ, Timonen M, Isohanni M. Cytokine abnormalities, inflammation and psychosis in the northern finland 1966 birth cohort. European Psychiatry 2014; 29: S519.
- [Background] Miller BJ, Dias JK, Lemos HP, Buckley PF. An open-label, pilot trial of adjunctive tocilizumab in schizophrenia. J Clin Psychiatry. 2016 Feb;77(2):275-6. doi: 10.4088/JCP.15l09920. No abstract available. PMID 26930525